CLINICAL TRIAL: NCT03914833
Title: Impact of Sports-related Concussions on the Attention and Executive Skills of Adolescents and Young Adults: Links With Subjective Symptoms and Recovery.
Acronym: EXAECOS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BEJOT 2018-2
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Sports-related Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Patients aged 13 to 25 years old with a concussion in sports practice less than 72 hours previously
  Interventions: Other: Questionnaires at inclusion, M1 and M3
- Control - High-level athelete: healthy subjects aged 13 to 25 years students at one of the partner institutions
  Interventions: Other: Inclusion Questionnaires
- Control - Non-high-level athelete: healthy subjects aged 13 to 25 years students at one of the partner institutions
  Interventions: Other: Inclusion Questionnaires

INTERVENTIONS:
Other: Inclusion Questionnaires — During the inclusion visit, neuropsychologist tests the scales: SCAT3 (Sport Concussion Assessment Test 3ème version), Trail-making test (TMT), Wechsler Adult Intelligence Scale (WAIS) TAP, HAS (Hospital Anxiety and Depression scale) ; PSQI (Pittsburg Sleep Quality Scale) ; RPQ (Rivermead Post concussion symptoms Questionnaire) ; and RHFUQ (Rivermead head injury follow-up questionnaire)
  Groups: Control - High-level athelete; Control - Non-high-level athelete
Other: Questionnaires at inclusion, M1 and M3 — During the inclusion visit, the 1-month visit and the 3-month visit; neuropsychologist grading of the scales: SCAT3 (Sport Concussion Assessment Test 3ème version), Trail-making test (TMT), Wechsler Adult Intelligence Scale (WAIS) TAP, HAS (Hospital Anxiety and Depression scale) ; PSQI (Pittsburg Sleep Quality Index) ; RPQ (Rivermead Post concussion symptoms Questionnaire) ; and RHFUQ (Rivermead head injury follow-up questionnaire)
  Groups: Patients

SUMMARY:
Concussion in sports ("Sports-Related Concussion" or "SRC") are a public health issue. The management of these injuries is evolving rapidly and decisions to return to play are based on clinical judgment. It is now recognized that the assessment of cognitive function must be one of the components of the assessment, in particular, in the protocol used to decide if a patient can resume practice. The available scales include only a brief cognitive assessment but do not provide an understanding of the level of deficit treatment. The use of computerized TAP (Test of Attentionnal Performance) tests, including finer measures of reaction time and apprehending the different attention and executive components (alertnes, orientation, flexibility, inhibition, updating), would allow a better understanding of the nature of the disorder and link it to subjective symptoms, and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given his non-opposition
* For minor controls: Written authorization and non-opposition from the 2 holders of parental authority beforehand.
* For minor patients: non-opposition from the 2 holders of parental authority
* For patients: patients aged 13 to 25 years old who have suffered a concussion in sports practice less than 72 hours previously and who consult at the CMRR of the CHU Dijon Bourgogne
* For controls: healthy subjects aged 13 to 25 years old students in one of the partner schools (Lycée les Arcades de Dijon, Lycée Saint Joseph, Dijon; Collège Marcel Pardé, Dijon; CREPS (Centre de Ressources et d'Expertise à la Performance Sportive) who have not had a concussion.

Exclusion Criteria:

* Person subject to legal protection (curatorship, guardianship)
* Person subject to limited judicial protection
* Pregnant, parturient or breastfeeding woman
* Major unable to consent
* For controls: subjects with a history of learning disabilities and/or concussion (identification of this history on the SCAT3 inclusion questionnaire).

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients consulting at the CMRR of the CHU Dijon Bourgogne
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Reaction time on the TAP computerized battery | Through study completion, an average of 23 month
Number of errors on the TAP computerized battery | Through study completion, an average of 23 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France